CLINICAL TRIAL: NCT00290992
Title: Open-Label, Multi-Center Study of SR29142 as Uricolytic Therapy/Prophylaxis for Hyperuricemia in Pediatric Patients With Newly Diagnosed Hematological Malignancies at High Risk for Tumor Lysis Syndrome
Brief Title: Rasburicase for Hyperuricemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study director, sanofi-aventis
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT5080
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: urate oxidase, hyperuricemia, lymphoma, leukemia
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Hyperuricemia; Lymphoma; Leukemia | interventions — rasburicase; Urate Oxidase

INTERVENTIONS:
Drug: rasburicase (SR29142)

SUMMARY:
Primary: To estimate efficacy of SR29142 to the pediatric patients with newly diagnosed hematological malignancies at high risk for Tumor Lysis Syndrome, by evaluation of plasma uric acid concentration.

Secondary: To investigate the safety in this population and anti-SR29142 antibodies, anti-SCP antibodies, and pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* <18 years of age
* Patient with newly diagnosed hematological malignancies presenting with hyperuricemia:
* Uric acid > 7.5 mg/dL in patients ≥ 13 years old- Uric acid > 6.5mg/dL in patients <13 years old

Or, patient with newly diagnosed hematological malignancies presenting with high tumor burden defined:

* Non-Hodgkin's lymphoma, Stage IV regardless of uric acid level,
* Non-Hodgkin's Lymphomas stage III regardless of uric acid level with one of the following:

  * At least one lymph node or mass >5 cm in diameter
  * LDH ≥ 3 x ULN (IU/L): Judging according to modified Murphy's classification
* Acute leukemia with white blood cell count (WBC) ≥ 50,000/mm3 or LDH ≥ 3 x ULN (IU/L) regardless of uric acid level. etc.

Exclusion Criteria:

* Patients who have received or are scheduled to receive other investigational drugs in 30 days prior to the start of SR29142 administration or during the trial period.
* Low birth weight infant (<2500g) or gestational age <37 weeks
* Patients who have received or are scheduled allopurinol within 72 hrs prior to the first dose of SR29142 or during the trial period.
* Known history of severe allergic reaction and/or severe asthma.
* Known history or family history of glucose-6-phosphate dehydrogenase deficiency.
* Known history of hemolysis and methemoglobinemia.
* Severe disorders of liver or kidney. ALT (GPT) > 5.0 x ULN, Total Bilirubin > 3.0 x ULN, Creatinine > 3.0 x ULN
* Uncontrollable infections (including viral infections).
* Known positive tests for HBs antigen, HCV antibodies, or HIV-1, 2 antibodies. etc.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Patients with a plasma uric acid level decreased to the endpoint by 48 hr after the start of first drug infusion and lasting until 24 hr after the start of final (Day 5) drug infusion.

SECONDARY OUTCOMES:
Safety will be assessed on clinical observation, laboratory test, vital sign (blood pressure, pulse rate and body temperature), and the occurrence of adverse events.
G6PD activity will be measured in only patients who demonstrate hemolysis.
Anti-SR29142 antibody and Anti-SCP antibody will be measured.
PK parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Keiji OHNO, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan